CLINICAL TRIAL: NCT02969967
Title: Effectiveness of a Dynamic Wrist-hand Orthosis in Early Outpatient Rehabilitation of the Upper Extremity Post Stroke: a Multiple Single Subject Design Evaluation
Brief Title: Effectiveness of a Dynamic Wrist-hand Orthosis in Early Outpatient Rehabilitation of the Upper Extremity Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2016:285
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2016-11

CONDITIONS: Stroke
Keywords: rehabilitation; upper extremity; orthosis; SaeboFlex
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SaeboFlex (Experimental): Use of the SaeboFlex orthosis for a set protocol of grasp-release activities
  Interventions: Device: SaeboFlex

INTERVENTIONS:
Device: SaeboFlex — Use of the SaeboFlex orthosis for a set protocol of grasp-release activities for 50 minutes at least 3 times per week, followed by 10 minutes of grasp-release activities without the orthosis for 8 weeks. Will occur in participants' homes after discharge from inpatient rehabilitation with visit from principal investigator to progress program for 1 hour 3 times a week for the first 2 weeks and then once a week for 6 weeks.
  Other Names: functional dynamic orthosis

SUMMARY:
The purpose of this study is to explore the effectiveness of the SaeboFlex orthosis in improving upper extremity recovery for people in the early phases of rehabilitation post stroke. The objectives of the study are:

1. to explore the effectiveness of the SaeboFlex orthosis in improving upper extremity function, strength, movement, spasticity and self-perceived occupational performance, in addition to conventional therapy, with continued use immediately after discharge from inpatient stroke rehabilitation and while waiting for outpatient occupational therapy services
2. to explore the relationship between the participants' level of self-efficacy and use of the SaeboFlex orthosis in the home environment
3. to explore the participants' experience of use of the SaeboFlex orthosis in the home environment.

DETAILED DESCRIPTION:
Although intensive and repetitive use of the paretic upper extremity has been shown to improve upper extremity outcomes post stroke, few therapeutic approaches allow those with moderate to severe upper extremity impairment to independently participate in repetitive grasp and release activities. The SaeboFlex orthosis is a dynamic wrist-hand orthosis that assists with finger and thumb extension after functional grasping with the paretic hand and therefore may allow those with more affected upper extremities post stroke to participate in repetitive grasp and release activities that they otherwise would be unable to do. More research is required on the effectiveness of this orthosis in improving upper extremity recovery post stroke especially when used at home as a continuation of therapy received during inpatient rehabilitation. It has been suggested that guided home rehabilitation programs can improve the ability of stroke survivors to be more independent in their activities of daily living. This study is a mixed methods study combining a quantitative single subject ABA design and qualitative post study individual interviews to first capture quantitative information on the effectiveness of the SaeboFlex intervention and then qualitative information that will build on and further explain the quantitative data. Three participants who are using a SaeboFlex orthosis as part of their upper extremity rehabilitation program will be recruited from an inpatient stroke rehabilitation unit as they are being discharged from inpatient rehabilitation and will be seen by the principal investigator in their homes for 1 hour 3 times a week for 2 weeks and then once a week for 6 weeks while they are on the waiting list for outpatient occupational therapy services. The intervention will follow a set protocol of grasp-release activities using the SaeboFlex orthosis for 50 minutes at least 3 times per week, followed by 10 minutes of grasp-release activities without the orthosis, both of which will be graded to provide optimal upper extremity challenge throughout the intervention period. Repeated baseline assessments will be completed by a trained research assistant, in the participants' homes, within one week of discharge from inpatient stroke rehabilitation and will be repeated after 4 and 8 weeks of intervention, followed by individual interviews in the participants' homes.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 or over who have had a first stroke within the past 6 months
* admitted to Riverview Health Centre (Winnipeg, Canada) for stroke rehabilitation and are being discharged to home locations within the city of Winnipeg
* fit with and started using a custom SaeboFlex orthosis as an inpatient at Riverview Health Centre after having met the active and passive movement criteria required to use the SaeboFlex orthosis
* referred to outpatient Occupational Therapy at the Health Sciences Centre (Winnipeg, Canada) for ongoing upper extremity rehabilitation using a SaeboFlex orthosis
* able to commit to the time requirements of the study
* have a premorbid fully functional upper extremity
* able to speak and understand English
* able to follow multistep commands and understand the purpose and required use of the orthosis
* able to stand for at least 10 minutes
* have 3 times per week access to a caregiver to assist with donning the orthosis at home if required

Exclusion Criteria:

* Chedoke McMaster Stroke Assessment, Impairment Inventory (Shoulder Pain section) score of 1-3
* score of 3 or more on the Modified Ashworth Scale for elbow, wrist or finger flexors
* swan neck deformities or contractures of the fingers or wrist of the paretic upper extremity
* history of skin breakdown on the paretic upper extremity or a score of less than 6 out of 12 on the Sensation Section of the Fugl-Meyer Upper Extremity Assessment
* significant cognitive impairment as determined by a score of 21 or less on the Montreal Cognitive Assessment
* able to fully extend fingers 10 times in a position of maximal shoulder flexion and elbow extension with a neutral wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Arm Activity Measure (ArmA) | Change from baseline upper extremity function to 4 and 8 weeks
  The Arm Activity Measure (ArmA) is a self-report tool designed for use with upper extremity spasticity management interventions. The ArmA was chosen because it provides a comprehensive assessment at the activity level of both active and passive upper extremity function; it is comprised of an 8 item passive function subscale and a 13 item active function subscale. Both subscales have been found to have high internal consistency and test-retest reliability.
Chedoke Arm and Hand Activity Inventory-7 (CAHAI-7) | Change from baseline upper extremity function to 4 and 8 weeks
  The Chedoke Arm and Hand Activity Inventory-7 (CAHAI-7) is a commonly used upper extremity functional assessment post stroke. It is comprised of seven bilateral functional tasks and has been found to have excellent test-retest and inter-rater reliability as well as internal consistency.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment-Upper Extremity (FMA-UE) | Change from baseline upper extremity impairment to 4 and 8 weeks
  The Fugl-Meyer Assessment-Upper Extremity (FMA-UE) is a widely used measure of motor impairment post stroke and is comprised of 33 items related to upper extremity movement. The FMA-UE has excellent inter-rater and test-retest reliability as well as construct validity in persons with stroke.
Stroke Impact Scale (SIS) | Change from baseline perception of recovery to 4 and 8 weeks
  The Stroke Impact Scale (SIS) is a well known and well studied measure of stroke survivors' perception of their recovery post stroke. The SIS has been widely used in stroke intervention studies.
Modified Ashworth Scale (MAS) | Change from baseline spasticity to 4 and 8 weeks
  The Modified Ashworth Scale (MAS) is a well known measure of spasticity post stroke. The MAS assesses the resistance to passive muscle stretch and is graded on a 6 point ordinal scale. The participants' elbow, wrist and finger flexors will be assessed with the MAS.
Hand Grip Strength (measured using dynamometry) | Change from baseline grip strength to 4 and 8 weeks
  Measurement of hand grip strength using dynamometry is common post stroke and has excellent test-retest and inter-rater reliability. An average of 3 grip strength trials will be taken at each measurement point using dynamometry.
Stroke Self-Efficacy Questionnaire (SSEQ) | Change from baseline self-efficacy to 4 and 8 weeks
  The Stroke Self-Efficacy Questionnaire (SSEQ) was designed to assess self-efficacy related to functional performance and self-management post stroke. The SSEQ is comprised of two subscales that are scored separately and correlate strongly with other measures of self-efficacy post stroke.
Canadian Occupational Performance Measure (COPM) | Change from baseline perception of occupational performance to 4 and 8 weeks
  The Canadian Occupational Performance Measure (COPM) is a valid and responsive measure of occupational performance and has been widely used in stroke research. The COPM uses a semi-structured interview format where performance and satisfaction scores will be identified for the participants' self-identified occupational performance issues.

OTHER OUTCOMES:
Individual interviews | 8 weeks
  Individual interviews will be conducted at 8 weeks, after the intervention is complete, to generate discussion about the perceived usability of the SaeboFlex orthosis in the home environment, the perceived effect on upper extremity recovery as well as the perceived relationship between self-efficacy and use of the SaeboFlex orthosis in the home environment.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda L Semenko, BMR (OT), Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birkenmeier RL, Prager EM, Lang CE. Translating animal doses of task-specific training to people with chronic stroke in 1-hour therapy sessions: a proof-of-concept study. Neurorehabil Neural Repair. 2010 Sep;24(7):620-35. doi: 10.1177/1545968310361957. Epub 2010 Apr 27. PMID 20424192
- [Background] Waddell KJ, Birkenmeier RL, Moore JL, Hornby TG, Lang CE. Feasibility of high-repetition, task-specific training for individuals with upper-extremity paresis. Am J Occup Ther. 2014 Jul-Aug;68(4):444-53. doi: 10.5014/ajot.2014.011619. PMID 25005508
- [Background] Butler A, Blanton S, Rowe V, Wolf S. Attempting to improve function and quality of life using the FTM Protocol: case report. J Neurol Phys Ther. 2006 Sep;30(3):148-56. doi: 10.1097/01.npt.0000281952.93934.6b. PMID 17029658
- [Background] Legg L, Langhorne P; Outpatient Service Trialists. Rehabilitation therapy services for stroke patients living at home: systematic review of randomised trials. Lancet. 2004 Jan 31;363(9406):352-6. doi: 10.1016/S0140-6736(04)15434-2. PMID 15070563